CLINICAL TRIAL: NCT00495781
Title: Swiss Functional Iron Deficiency Study
Brief Title: Out Come Study To Define Laboratory Parameters That Are Best Suited to Diagnose Functional Iron Deficiency
Acronym: SFIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spital Zollikerberg (Other)
Collaborators: Viollier Inc. (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SFIDS-2004
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2007-07-03 (Estimated); Status verified 2007-07

CONDITIONS: Functional Iron Deficiency
Keywords: functional iron deficiency; renal anemia; dialysis; erythropoietin; darbepoetin
MeSH Terms: interventions — Peroxisomal Biogenesis Factor 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: %-hypo (laboratory parameter, functional iron deficiency)
Procedure: CHr (laboratory parameter, functional iron deficiency)
Procedure: RET-HE (laboratory parameter, functional iron deficiency)

SUMMARY:
The purpose of the study is to define laboratory parameters which are best suited to diagnose functional iron deficiency. Functional iron deficiency is a condition where - due to the lack of iron bioavailability - the patient suffers from symptoms such as fatigue and weakness, or his/her capacity to produce red blood cells is reduced.

DETAILED DESCRIPTION:
In dialysis patients the degree of anemia is highly correlated to both morbidity and mortality. A drop in Hb by 10 g/L translates into an increase in the rate of hospitalizations of 5 to 6 % and a rise in mortality by 4 to 5 %. The past two decades have seen great progress in the treatment of renal anemia with the advent of erythropoietin, and, more recently, darbepoetin. Quite soon, however, it became clear, that anemia in patients with chronic renal failure is complicated by a lack of bioavailable iron, which confers these patients partly resistant to treatment with erythropoietin/darbepoetin.

There are several parameters in use to estimate total body iron stores in the diagnosis of iron deficiency and iron deficiency anemia. Serum iron represents only a minor fraction of total body iron and is subject to major fluctuations due to influx or efflux from tissue iron stores. In addition, it shows a great diurnal variability, and is therefore a very poor parameter of iron deficiency. Iron saturation of its transporter protein in blood, transferrin, is similarly difficult to interpret, as it depends also in part on the determination of serum iron levels. Ferritin, the tissue iron storage protein, is released into the circulation during active liver cell damage, and, quite unlike serum transferrin levels, ferritin levels rise during the acute phase response of the inflammatory reaction. In most cases, however, the serum ferritin level, if substantiated by the concurrent determination of the C-reactive protein and the alanine-leucine-aminotransferase (ALT) to exclude both, occult liver cell damage and inflammation, correlates well with total body iron stores and total body iron deficiency, respectively.

The serum ferritin level, however, is a poor marker of functional iron deficiency when erythropoiesis is inhibited by the relative lack bioavailable iron in high turnover states of the bone marrow such as in hemolysis and in the thalassemias. Correspondingly, in patients with hemochromatosis and an increased functional iron availability, erythropoiesis will be augmented following acute blood losses.

To date no golden standard exists to measure functional iron deficiency in a routine clinical setting. As a matter of fact, in some clinical studies functional iron deficiency is still diagnosed indirectly and retrospectively by the effect of an iron substitution therapy (increase in Hb by 10 g/L following 4 weeks of iron supplementation)

The percentage of hemoglobin-deficient, hypochromic erythrocytes, as measured by some hemocytometers, reflects the availability of iron for erythropoiesis and has become a surrogate marker of functional iron deficiency. As the lifespan of erythrocytes varies according to the degree of the patient's uremia between approximately 60 and 120 days, hypochromic erythrocytes, measured as a percentage of total erythrocytes (%-Hypo), become detectable only late in the course of erythropoietin therapy, and are therefore thought by some to be of only limited sensitivity in the diagnosis of functional iron deficiency.

With the automated measurement of reticulocytes, it has become now possible on some hemocytometers, such as the Advia 120, to also determine the hemoglobin content in newly formed reticulocytes (CHr). The hemoglobin content of reticulocytes mirrors more closely the current availability of iron for erythropoiesis. What would make CHr so attractive for clinicians and the clinical laboratory, is not only its acclaimed sensitivity to detect functional iron deficiency, but, even more so, its easy availability, as it forms part of a simple reticulocyte count on a normal hemocytometer.

In other hemocytometric systems laser light scatter patterns have been utilized to characterize the hemoglobin content in reticulocytes (RET-HE). This new parameter, RET-HE, has been shown to be of a similar sensitivity and specificity as CHr and to give comparable results in clinical samples (CHr, r = 0.94).

The present study is meant to define the laboratory parameter (%-Hypo/CHr or RET-He) which is suited best to diagnose functional iron deficiency. The study design asks for the parameter with which physicians will be able to diagnose their patients so to improve the management of their anemia. A diagnostic parameter is searched for which improves the patients' treatment the most, as measured by blood hemoglobin levels (primary end point 1), at the lowest possible costs (primary end point 2).

ELIGIBILITY:
Inclusion Criteria:

* renal anemia, glomerular filtration rate < 10 ml/min
* therapy with either erythropoietin or darbepoetin
* dialysis patients
* therapy with iron

Exclusion Criteria:

* cancer
* autoimmune diseases
* chronic inflammation
* liver disease
* thalassemia, and other causes of anemia (except for renal anemia and iron deficiency anemia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2004-10; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin | 12 months
Costs = erythropoietin/darbepoetin prescribed | 12 months

SECONDARY OUTCOMES:
Changes in soluble transferrin receptor | 12 months
Changes in transferrin saturation | 12 months
changes in ferritin | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Boris E Schleifenbaum, MD, Principal Investigator — Viollier Inc.
Locations (1):
- Spital Zollikerberg, Zollikerberg, Canton of Zurich, Switzerland